CLINICAL TRIAL: NCT05887284
Title: Investigation of the Clinical Efficacy of Low-dose Ionizing Radiation in the Treatment of Osteoarthritis
Acronym: IMMO-LDRT02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IMMO-LDRT02
Record Dates: First submitted 2023-05-05; First posted 2023-06-02 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Arthrosis; Osteoarthritis
Keywords: low dose radiotherapy; LDRT
MeSH Terms: conditions — Osteoarthritis | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose Radiation Therapy (Experimental): In the test group, patients receive radiotherapy with six fractions of 0.5 Gy each over a period of 3 weeks, with 2 doses applied per week (total dose 3.0 Gy). After the 1st follow-up (3 months after radiotherapy), patients receive the patients in both arms have the option to receive a 2nd series of radiotherapy in consultation with the study physician if no improvement in symptoms has occurred or patients are still not sufficiently satisfied with the outcome (this decision is still made by the physician and patient in a blinded manner). The patients from the test group receive another irradiation series with six fractions of 0.5 Gy each according to the same schedule as before (total dose 3.0 Gy and in sum with the first series 6.0 Gy).
  Interventions: Radiation: low dose radiotherapy (0.5 Gy)
- Mock Radiation Therapy (Placebo Comparator): In the control group, patients receive sham irradiation with six fractions of 0.0 Gy each over a period of 3 weeks, with 2 treatments per week. After the 1st follow-up (3 months after radiotherapy), patients receive the patients in both arms have the option to receive a 2nd series of radiotherapy in consultation with the study physician if no improvement in symptoms has occurred or patients are still not sufficiently satisfied with the outcome (this decision is still made by the physician and patient in a blinded manner). The patients in the control group, on the other hand, now also receive a radiotherapy with six fractions of 1.0 Gy each over a period of 3 weeks with 2 fractions per week (total dose 6.0 Gy).
  Interventions: Radiation: mock radiation treatment; Radiation: low dose radiotherapy (1.0 Gy)

INTERVENTIONS:
Radiation: low dose radiotherapy (0.5 Gy) — 12 times 0.5 Gy
  Arms: Low dose Radiation Therapy
Radiation: mock radiation treatment — 6 times 0.0 Gy
  Arms: Mock Radiation Therapy
Radiation: low dose radiotherapy (1.0 Gy) — 6 times 1.0 Gy
  Arms: Mock Radiation Therapy

SUMMARY:
IMMO-LDRT02 is a prospective, placebo-controlled, double-blind, randomized trial to investigate the clinical efficacy of low dose radiation therapy (LDRT) in the treatment of arthrosis. Newly diagnosed or already existing arthroses of the fingers, wrists, shoulders, knees, ankles and feet will be enclosed. Finally, the evidence of clinical benefit from LDRT (6 x 0.5 Gy) will be compared to the placebo group (6 x 0 Gy), by determination via a visual analog scale and identification of immunological changes.

DETAILED DESCRIPTION:
The prevalence of chronic degenerative and inflammatory disorders, such as osteoarthritis, is constantly rising. As not all patients do respond adequately to the standard therapies, alternative treatment options such as low dose radiation therapy (LDRT) has gained further importance. LDRT is known to induce a long-lasting pain reduction, while having few side effects. Nonetheless, the detailed biological and immunological modes of action remain mostly elusive. In addition, there is a lack in placebo controlled randomised controlled trials (RCTs) proofing the pain-relieving effects of LDRT. So, the prospective, placebo-controlled, double-blind, randomized IMMO-LDRT02 trial to investigate the clinical efficacy of LDRT in the treatment of arthrosis should close this gap. Newly diagnosed or already existing arthroses of the fingers, wrists, shoulders, knees, ankles and feet will be enclosed. Finally, the evidence of clinical benefit from LDRT (6 x 0.5 Gy) will be compared to the placebo group (6 x 0 Gy), by determination via a visual analog scale (VAS) and identification of immunological changes, which contribute to the success of therapy and are specifically found in the test group (IMMO-LDRT01 trial; ClinicalTrials.gov Identifier: NCT02653079).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed osteoarthritis according to ACR criteria (exclusion of other other arthritides and chronic rheumatoid arthritis via laboratory tests):

  * Finger and wrist osteoarthritis
  * Elbow arthrosis
  * Shoulder arthrosis
  * Knee arthrosis
  * Ankle and foot joint arthrosis
* First time application of low-dose radiotherapy (LDRT) of the affected joint.
* Willingness to cooperate and accessibility of the patients (geographical proximity) for treatment and Follow-up care

Exclusion Criteria:

* Patients with tumor diseases
* People capable of childbearing or procreation who do not take consistent contraceptive measures during therapy
* Persistent drug, medication or alcohol abuse
* Patients for whom, in the physician's judgment, participation is not justifiable with regard to their well-being due to temporary withdrawal of standard medication.
* Patients in whom the diagnosis of osteoarthritis of the affected joint cannot be made without doubt. To establish the diagnosis, the guidelines of the American College of Rheumatology (ACR) are followed.
* Earlier radiation therapy for treatment of cancer

Min Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in general pain (determined by visual analog scale (VAS) score) after LDRT compared to the placebo. | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  Determination of the general pain level by determining a so-called pain score which is calculated from the parameters pain level (VAS) and pain history (duration, frequency, maximum, quality and occurrence of pain). VAS is determined from 0 (no pain) to 10 (maximum pain). Pain history will also assessed bei an scale from 1 to 10.
Identification of immunological changes, which contribute to the success of therapy and are specifically found in the test group. | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  Longitudinal Immunophenotyping of the patients: Detection of about 30 distinct immune cell (sub)types together with their activation markers during treatment.

SECONDARY OUTCOMES:
Evidence of an objectionable clinical benefit of LDRT for finger/wrist osteoarthritis. | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  Analysis of the pain-free finger and hand force by using finger and hand strength meter.
Analysis of the efficacy of LDRT against placebo in modulating patient's well-being. | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  Determination of disease activity and pain using the international accepted EuroQol Research Foundation questionnaire EQ-5D-5L (IMMOLDRT02/EQ-5D-5L). Scale of EQ-5D-5L is from 5 (perfect well being) to 25 (illness with pain).
Analysis of the clinical efficacy of LDRT against placebo in fingers / wrists. | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  Determination of disease activity and pain in treated Fingers / Wrists using international disease specific questionnaires (AUSCAN score). Scaled on 5-point Likert, 100mm Visual Analog and 11-box Numerical Rating Scales, the AUSCAN™ 3.1 is a valid, reliable and responsive measure of outcome. Scale from 0 (no pain) to 100 (worst pain).
Analysis of the clinical efficacy of LDRT against placebo in shoulders. | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  Determination of disease activity and pain in treated shoulders using international disease specific questionnaires (Oxford Shoulder Questionnaire (OSS). Score from 12 (no trouble) to 60 impossible to do).
Analysis of the clinical efficacy of LDRT against placebo in knees. | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  Determination of disease activity and pain in treated knees using international disease specific questionnaires (Oxford Knee Questionnaire). Score from 12 (no trouble) to 60 impossible to do).
Analysis of the clinical efficacy of LDRT against placebo in foot and ankle joints. | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  Determination of disease activity and pain in treated foot and ankle joints using international disease specific questionnaires (EFAS European Foot and ankle score questionnaire). Score from 0 (no problems) to 40 impossible to do).
Documentation and examination of general medication and pain medication. | From Randomisation (day 0) till end of the trial (day 336), assessed every 7 days from day 0 to day 336..
  Collection of patient's drug use by electronic medication diary.
Investigation of the drop-out rate in the test and control group. | Fraom day of randomisation (day 0) till patient's independent trial abort or day 336, whichever came first.
  Determination of the patients number changing the group from placebo to treatment group.
Comparison of the two series with single doses 0.5 Gy against one series with single dose 1.0 Gy with regard to pain score reduction and immunological changes | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  Determination of the general pain level by determining a so-called pain score which is calculated from the parameters pain level (VAS) and pain history (duration, frequency, maximum, quality and occurrence of pain). VAS is determined from 0 (no pain) to 10 (maximum pain). Pain history will also assessed bei an scale from 1 to 10.
Modulation-matrix of immune cell function. | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  After blood collection, immune cells were separated and harvested. Cells are differentiated ex-vivo into mature immune cell sub populations, and their functionality is assessed by staining with surface markers using multicolour flowcytometry. Functionality is described by the amount of differentiable cells.
Detection of chromosome aberrations | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  After blood collection, the immune cells were separated and harvested. The cells are examined ex-vivo for the occurrence of chromosomal aberrations using the multicolour Fluorescence in situ hybridization (FISH) method. The number of chromosomal defects as well as the type is recorded. Comparison is then made with normal human donors as well as the between study groups.
Investigation of side effect profile of LDRT | Day 0 till end of the trial at the distinct time points of end of first LDRT series (day 28), first follow up (day 112), end of second LDRT series (day 140), second follow up (day 224), final follow up (day336).
  The adverse effects of LDRT is recorded by official questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Ott, Prof. Dr, Study Director — Department of Radiation Oncology, Uniklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg; Benjamin Frey, PD Dr.-Ing., Principal Investigator — Translational Radiobiology, Department of Radiation Oncology, Uniklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg; Thomas Weissmann, Dr., Principal Investigator — Department of Radiation Oncology, Uniklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg; Rainer Fietkau, Prof. Dr., Study Chair — Department of Radiation Oncology, Uniklinikum Erlangen, Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- Department of Radiation Oncology, Universitätsklinikum Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No